CLINICAL TRIAL: NCT01683630
Title: Comparison of the Epidemiology and Clinical Outcomes of Laboratory-Confirmed Influenza A and Influenza B Cases in Manitoba, Canada
Brief Title: Comparison of Epidemiology and Clinical Outcomes of Influenza A & B Cases in Manitoba, Canada
Status: Completed | Type: Observational
Sponsor: International Centre for Infectious Diseases, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: ICID-2012-FLU-A,B-02
Record Dates: First submitted 2012-08-31; First posted 2012-09-12 (Estimated); Results first posted 2015-10-19 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Influenza; Influenza type A; Influenza type B; hospitalization; Manitoba; Canada
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Confirmed influenza A and B cases: Cases of influenza A and B as diagnosed by PCR, viral culture or florescence microscopy

SUMMARY:
This study compares the epidemiology and clinical outcomes of laboratory confirmed influenza type A to type B following clinical diagnosis of influenza. Multivariate models are used to assess the effects of influenza type on clinical outcomes while accounting for potential confounders.

DETAILED DESCRIPTION:
Annual epidemics of influenza are an important public health problem globally and in Canada. Each year, 10-25% of the Canadian population become infected with influenza. Most of these infections are typically asymptomatic or associated with a mild self-limiting illness. However, influenza can cause severe illness leading to hospitalization and death, especially among the very young, the elderly and among those with underlying chronic conditions. It has been estimated that on average about 4,000 influenza-related deaths occur in Canada each year. In addition, the economic burden of influenza is significant because of the high direct costs associated with increased utilization of services and the indirect costs caused by school and work absenteeism.

This project compares laboratory-confirmed cases of influenza A and B in terms of their epidemiology, and the overall and cause-specific incidence rates of important clinical outcomes including physician visits, hospitalization and death following clinical diagnosis of influenza cases in Manitoba over the period from 1993 to 2008.

The study assesses secular and seasonal trends in the incidence rates of influenza A and B cases in Manitoba during the period of 1993-2008, to determine whether these rates vary for different subsets of the population defined by demographic (e.g., age group, gender), socioeconomic, geographic (neighborhood of residence) and clinical (e.g., vaccination, presence of chronic conditions, immune status) characteristics.

The analysis by influenza type then compares the overall and cause-specific incidence rates of physician visits, hospitalization and death following the diagnosis of a laboratory-confirmed influenza. The effects of influenza type on clinical outcomes (e.g., hospitalization) are assessed with multivariate models while accounting for potential confounding by demographic, socioeconomic, geographic and clinical (e.g., co-morbidity, immune status) characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Any person who normally resides in Manitoba and who has been continuously covered by Manitoba Health during the study period will be eligible for inclusion in the study.

Exclusion Criteria:

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person who normally resides in Manitoba and who has been continuously covered during the study period will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1849 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salah Mahmud, MD, PhD, Principal Investigator — Associate Professor, University of Manitoba
Locations (1):
- International Centre for Infectious Diseases, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hinds AM, Bozat-Emre S, Van Caeseele P, Mahmud SM. Comparison of the epidemiology of laboratory-confirmed influenza A and influenza B cases in Manitoba, Canada. BMC Public Health. 2015 Jan 30;15:35. doi: 10.1186/s12889-015-1351-z. PMID 25633280

RESULTS

PARTICIPANT FLOW:
Groups:
- Confirmed Cases of Influenza A: Laboratory confirmed cases of influenza A diagnosed by PCR, viral culture or florescence microscopy
- Confirmed Cases of Influenza B: Laboratory confirmed cases of influenza B diagnosed by PCR, viral culture or florescence microscopy
Period: Overall Study
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B
Started | 1404 | 445
Completed | 1404 | 445
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B | Total
Number analyzed (Participants) | 1404 | 445 | 1849
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 511 | 236 | 747
  Between 18 and 65 years | 325 | 129 | 454
  >=65 years | 568 | 80 | 648
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 758 | 245 | 1003
  Male | 646 | 200 | 846
Region of Enrollment [Number; unit: participants]
  Canada | 1404 | 445 | 1849

OUTCOME MEASURES:

1. Primary Outcome: Age Adjusted Percentage of Participants With a Physician Visit Due to Any Diagnosis Within 30 Days of the Index Date of the Confirmed Influenza A and B Cases in the Province of Manitoba
Time Frame: up to 15 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B
Number analyzed (Participants) | 1404 | 445
Percentage of participants | 23.5 [22.2 to 24.8] | 22.1 [20.1 to 24.1]

2. Primary Outcome: Percentage of Participants With a Risk of Hospitalization Due to Any Diagnosis Within 30 Days Following the Index Date of Confirmed Cases of Influenza A and B in the Province of Manitoba
Time Frame: upto 15 years
Measure: Number; unit: Percentage of participants
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B
Number analyzed (Participants) | 1404 | 445
Percentage of participants | 9.0 | 7.0

3. Primary Outcome: Risk of Death Due to Any Cause During 30 Days Following the Index Date of Laboratory Confirmed Cases of Influenza A and B in the Province of Manitoba
Time Frame: Upto 15 years
Measure: Number; unit: percentage of participants
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B
Number analyzed (Participants) | 1404 | 445
percentage of participants | 4.5 | 2.0

ADVERSE EVENTS:
Time Frame: 0 months
Description: Serious and other Adverse Events were not collected/assessed
Arm/Group | Confirmed Cases of Influenza A | Confirmed Cases of Influenza B
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No